CLINICAL TRIAL: NCT00262392
Title: Study Into the Effect of Pamidronate for the Prevention of Heterotopic Ossification in High-risk Patients: A Randomized Controlled Trial
Brief Title: Study of Pamidronate for the Prevention of Heterotopic Ossification
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: FAG (Freie Medizinische Gesellschaft) (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PamidronateforHO271005; HO
Record Dates: First submitted 2005-12-05; First posted 2005-12-06 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2015-03

CONDITIONS: Heterotopic Ossification
Keywords: heterotopic ossification,; prevention,; high risk,; bisphosphonates,; radiotherapy
MeSH Terms: conditions — Ossification, Heterotopic | interventions — Pamidronate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pamidronate (Experimental): Pamidronate
  Interventions: Drug: Pamidronate (AREDIA)
- radiation (Active Comparator): radiation
  Interventions: Drug: Pamidronate (AREDIA)

INTERVENTIONS:
Drug: Pamidronate (AREDIA) — Pamidronate (AREDIA) vs radiation

SUMMARY:
The purpose of this study is to determine whether Bisphosphonates in comparison to radiation therapy are effective in the prophylaxis and treatment of heterotopic ossification in high risk patients.

DETAILED DESCRIPTION:
BACKGROUND: The acquired form of heterotopic ossification (HO) is the most common type of extraskeletal ossification and usually precipitated by a trauma such as total hip arthroplasty [THA] or spinal cord injury. After THA the incidence of HO is as high as 50%, but may reach up to 90% in high risk populations leading to severe functional impairment with ankylotic loss of joint mobility. Nonsteroidal anti-inflammatory drugs (NSAIDs) and external radiation have been used in preventing HO. Specifically, patients with surgical resection of HO at the hip have a high postoperative relapsing rate. Best results were observed after prophylactic radiation treatment with disease recurrence in 33-45% of patients. Data on the effect of bisphosphonates in the prevention of postoperative HO are scarce and mainly limited to the use of the first generation bisphosphonate etidronate. In a retrospective observational study we observed a marked beneficial effect of pamidronate infusions: none of the high risk patients with established HO undergoing surgical removal presented with disease recurrence.

AIM: We therefore aim to prospectively confirm our findings and to evaluate the efficacy of pamidronate for the prevention of recurrent HO after surgical removal of ipsilateral HO. Clinical, biochemical and radiological treatment outcome will be compared to standard clinical practice using preoperative external radiation.

ENDPOINTS: Primary endpoint is the radiological HO recurrence rate. Secondary endpoints are the clinical, functional and biochemical outcome (as assessed by several clinical and laboratory markers).

METHODS: This prospective, randomized trial will be carried out at the University Hospital in Basel/Buderholz in collaboration with the Orthopedic Clinic of the Swiss Paraplegic Centre in Nottwil. Patients who are admitted to the one of the participating orthopedic clinics for removal of HO at the hip will be included in the study. A total number of 40 consecutive patients will be recruited (recruitment phase 24 months) and randomized in a "bisphosphonate group", treated with peri- and postoperative pamidronate infusions (1.0 mg/kg/day for 3 days) and in a "radiation group", treated with external radiation with a single dose of 7 Gy within 24 hours prior to surgical intervention. Additionally, both groups will be treated with NSAIDs for 14 days.

EXPECTED RESULTS: We hypothesize that in treating patients at risk, therapy with pamidronate will be superior in reducing the recurrence rate of established HO as compared to external radiation after surgical resection.

SIGNIFICANCE: Because of the high prevalence in selected risk patients and significant morbidity of HO, this study will offer potential for improving the management of HO. Our study is targeting patients with high risk to develop HO were highly effective prevention is still lacking. Furthermore, a diagnostic marker to identify patients at risk to develop HO would optimize disease management and would allow for early, more successful treatment.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients with established HO (Brooker grade III-IV), hospitalized for resection of HO lesions

Exclusion criteria:

* Age <20 years
* Vitamin D deficiency (25OH-Vitamin D <30 ng/ml)
* Renal insufficiency (Clearance <50 ml/min)
* Intolerance of bisphosphonates
* Unable to provide informed consent

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2005-06; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
Primary endpoint is the radiological Heterotopic Ossification recurrence rate. | 6 month

SECONDARY OUTCOMES:
Secondary endpoints are the clinical, functional and biochemical outcome (as assessed by several clinical and laboratory markers). | 6 month

CONTACTS AND LOCATIONS:
Overall Officials: philipp schuetz, MD, Principal Investigator — University Hospital, Basel, Switzerland; Christian Meier, MD, Study Director — University Hospital in Basel

REFERENCES:
- [Background] Schuetz P, Mueller B, Christ-Crain M, Dick W, Haas H. Amino-bisphosphonates in heterotopic ossification: first experience in five consecutive cases. Spinal Cord. 2005 Oct;43(10):604-10. doi: 10.1038/sj.sc.3101761. PMID 15867938